CLINICAL TRIAL: NCT00432406
Title: TNF-α Blockade for Psoriatic Arthritis - A Clinical and MRI Study, and the Effects on Cytokine and Cardiovascular Risk Profile
Brief Title: Tumor Necrosis Factors (TNF)-α Blockade for Psoriatic Arthritis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Edumun K Li, MD, The Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PSA-2006-002
Record Dates: First submitted 2007-02-06; First posted 2007-02-07 (Estimated); Last update posted 2009-03-11 (Estimated); Status verified 2009-03

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; TNF-α; Cardiovascular risk; Immunomodulatory activities
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — Infliximab; Etanercept

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): infliximab
  Interventions: Drug: Infliximab
- 2 (Active Comparator): etanercept
  Interventions: Drug: Etanercept

INTERVENTIONS:
Drug: Infliximab — Infliximab 5 mg/kg given at day 1, week 2, week 6
  Other Names: remicade
  Arms: 1
Drug: Etanercept — Etanercept 25 mg twice weekly
  Other Names: enbrel
  Arms: 2

SUMMARY:
The purpose of this study is:

* To elucidate the immunomodulating properties of anti-TNF-α therapy in patients with psoriatic arthritis (PsA).
* To ascertain whether magnetic resonance imaging (MRI) is a sensitive tool in measuring early response after therapy with anti-TNF-α in the PsA wrist using the Outcome Measures in Rheumatoid Arthritis Clinical Trials (OMERACT) guidelines for rheumatoid arthritis (RA).
* To assess whether the lipid and other cardiovascular risk profiles would improve after anti-TNF-α therapy in patients with PsA.

DETAILED DESCRIPTION:
The study was a 12-week, open-label trial of anti-TNF therapy in 20 consecutive patients (Group 1). Another 20 consecutive patients with active disease whom have met the exclusion criteria, or were unwilling to start anti-TNF therapy for fear of toxicity would be recruited as control patients (Group 2). 20 healthy controls were recruited for comparison of the metabolic risk factors (Group 3). Study visits for groups 1 and 2 were conducted at baseline, weeks 2 and 6, and then week 12.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or above
* PsA with active disease despite treatment with non-steroidal anti-inflammatory drug (NSAID)
* 3 or more swollen and tender joints
* Inadequate response after 4 weeks of, or intolerance to nonsteroidal anti-inflammatory drug therapy.
* Methotrexate (MTX) is allowed during the study only if it has been taken for at least 3 months previously, with the dosage stable for at least 4 weeks prior to the baseline visit.
* Prednisone ≤ 10 mg/day and/or nonsteroidal anti-inflammatory drugs must have been taken at stable dosage for at least 2 weeks before entering the trial.
* Informed consent

Exclusion Criteria:

* Little or no ability for self-care
* Used a DMARD other than methotrexate or received intra-articular, intramuscular, or intravenous corticosteroids in the 4 weeks before screening.
* Topical vitamin A (Neotigason CR) or D analog preparations (Daivonex CR), and anthralin for psoriasis within 2 weeks of baseline.
* Concurrent treatment with MTX at dosages > 15 mg/week and/or corticosteroids in a prednisone-equivalent dosage of > 10 mg/day.
* Prior anti-TNF therapy at any time.
* Infected joint prosthesis during the previous 5 years.
* Serious infections, such as hepatitis, pneumonia, pyelonephritis in the previous 3 months.
* Any chronic infectious disease such as renal infection, chest infection with bronchiectasis or sinusitis.
* Active tuberculosis requiring treatment within the previous 3 years.
* Opportunistic infections such as herpes zoster within the previous 2 months.
* Any evidence of active cytomegalovirus; active Pneumocystis carinii; or drug-resistant atypical mycobacterial infection.
* Known hypersensitivity to murine proteins
* Current signs or symptoms of severe, progressive, or uncontrolled renal, hepatic, haematological, gastrointestinal, endocrine, pulmonary, cardiac, neurological, or cerebral disease.
* A history of lymphoproliferative disease including lymphoma or signs suggestive of disease, such as lymphadenopathy of unusual size or location (ie, lymph nodes in the posterior triangle of the neck, infraclavicular epitrochlear, or periaortic areas); splenomegaly.
* Any known malignant disease except basal cell carcinoma currently or in the past 5 years.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2006-05; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Changes in the degree of inflammation as reflected by the MRI score, cytokines and chemokine levels | week 52
Changes in the cardiovascular risk factor levels which are directly mediated by TNF-α | week 52

SECONDARY OUTCOMES:
Number of patients who can achieve ACR 20 | week 52
Correlation of clinical parameter, inflammatory markers and MRI findings | week 52

CONTACTS AND LOCATIONS:
Overall Officials: Edmund K Li, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Prince of Wales Hospital, Hong Kong, China